CLINICAL TRIAL: NCT03433456
Title: Leveraging Ongoing Home Visitation Programs to Address Obesity Disparities Among Underserved, Low-Income Mothers and Children
Brief Title: Healthy Homes, Healthy Habits
Acronym: HABITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 000517527; 2U54MD000502-15 (NIH)
Record Dates: First submitted 2018-01-31; First posted 2018-02-14 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Obesity, Childhood; Obesity; Familial
Keywords: obesity; low-income; health disparities; home visitation; prevention; childhood obesity; habit
MeSH Terms: conditions — Obesity; Pediatric Obesity; Habits

STUDY DESIGN:
Intervention Model Description: Caregiver-child dyads will be randomized to either the intervention group (receiving home intervention + HABITS program) or the a control group to receive their standard of care (home intervention without HABITS)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home visitation + HABITS Program (Experimental): The HABITS module will target 5 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, decreasing fried foods, and encouraging regular self-monitoring and self-weighing) aimed at reducing obesity risk in mothers or primary caregivers and children. Participants will receive the HABITS module in addition to their standard home visitation services.
  Interventions: Behavioral: Home visitation + HABITS program; Behavioral: Standard home visitation program
- Standard home visitation program (Active Comparator): Participants will receive the standard of care home visitation regularly delivered through the existing home visitation program without the HABITS module.
  Interventions: Behavioral: Standard home visitation program

INTERVENTIONS:
Behavioral: Home visitation + HABITS program — The HABITS program will target 5 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, decreasing fried foods, and encouraging regular self-monitoring and self-weighing) aimed at reducing obesity risk in mothers or primary caregivers and children.
  Arms: Home visitation + HABITS Program
Behavioral: Standard home visitation program — Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on promoting caregiver and child health by providing screenings and referrals, encouraging smoking cessation, promoting safe sleep practices, and strengthening children's school readiness and achievement, social/emotional and physical development.

SUMMARY:
The purpose of this study is to evaluate whether an intervention targeting healthy habit development reduces the risk and prevalence of obesity in low-income mothers and children. The study intends to evaluate whether the intervention, delivered in the context of home visitation services for low-income families, reduces weight gain and risk factors associated with parent and childhood obesity compared to those receiving standard home visitation services.

DETAILED DESCRIPTION:
Participants will be 140 mothers (>50% African American; 100% meet federal poverty level) and their children (n=140; 0-4yo at baseline) (total of N=140 mother-child dyads; i.e., 140 mothers + 140 children = 280 total participants) enrolled in our home visitation partner in central Alabama. Home visitors will be randomly assigned to deliver the home visitation curriculum with or without HABITS (an obesity prevention program targeting key eating and activity behaviors) as part of their monthly home visits for 12 months. Treatment sessions for standard of care or standard + HABITS arms will be facilitated by trained home visitors. If a mother or primary caregiver and her child are randomized to participate in the HABITS + Standard home visitation curriculum, they will receive ~15 minutes of information, activities, and assistance regarding the development of key behaviors relating to obesity prevention, which will be imbedded within the existing home visitation curriculum. The HABITS program will address habit-formation of four behaviors relevant to mothers or primary caregivers and children: (1) limit fried foods; (2) limit sugar-sweetened beverages (SSB); (3) increase daily steps; (4) increase fruits and vegetables. Additionally, mothers or primary caregivers will also practice habit formation focused on self-monitoring of weight and the four behaviors previously mentioned. Skill training will focus on habit formation and home environment modification conducive to the four behaviors.

Mothers or primary caregivers in the intervention group will be provided the HABITS + standard home visitation program for 12 months, while those in the control group will be provided the standard home visitation program during this time. Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on promoting caregiver and child health by providing screenings and referrals, encouraging smoking cessation, promoting safe sleep practices, and strengthening children's school readiness and achievement, social/emotional and physical development.

ELIGIBILITY:
Inclusion Criteria:

*Important: Mother (or caregiver) and child dyads are enrolled together. Both must meet inclusion criteria to participate.

Mothers or Primary Caregivers:

* Age 18-75 years of age
* Enrollment in First Teacher Home Visiting Program (First Teacher) through the Family Guidance Center of Alabama.
* Mother or primary caregiver of 0-4 year old child
* Generally Healthy

Children:

* 0-4 years of age at time of enrollment
* Parent or primary caregiver enrolled in First Teacher

Exclusion Criteria:

Mothers or primary caregivers:

* Currently enrolled in a diet and weight loss program, AND either a) significant weight loss of 10+ pounds in the last 6 months, OR b) unwilling to discontinue from current diet and weight loss program.

Children:

* Child has a history of a feeding or eating disorder

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J. Salvy, PhD, Principal Investigator — University of Alabama at Birmingham; Gareth R. Dutton, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
With the documented permission of the IRB, the PI may develop a transportable de-identified database, codebook, and mechanism by which data can be shared with qualified investigators. Interested investigators will be asked to complete a standardized request form stating the specific aims of the analyses, the analytic plan, available resources for completing the proposed project, proposed timeline, and goals (i.e., manuscripts, presentations, and/or grant applications). The PI and research team will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to complete the request, and whether data will be adequately protected and managed. If any of these issues are problematic, the PI and research team will attempt to negotiate a fair resolution with the interested investigators and NIMHD program staff.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Background] Salvy SJ, Dutton GR, Borgatti A, Kim YI. Habit formation intervention to prevent obesity in low-income preschoolers and their mothers: A randomized controlled trial protocol. Contemp Clin Trials. 2018 Jul;70:88-98. doi: 10.1016/j.cct.2018.05.015. Epub 2018 May 24. PMID 29802965

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Started (This is the total number of caregivers and children who started the study.) | 158 | 138
Caregivers Started (Number of caregivers only who started the study.) | 79 | 69
Children Started (Number of children only who started the study.) | 79 | 69
Caregivers Completed (Number of caregivers only who completed the study.) | 71 | 63
Children Completed (Number of children only who completed the study.) | 71 | 63
Completed (This is the total number of caregivers and children who completed the study.) | 142 | 126
Not Completed | 16 | 12
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 14 | 11
Not completed — Pt in ICU and unable to complete follow-up visit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program | Total
Number analyzed (Participants) | 158 | 138 | 296
Age, Categorical [Count of Participants; unit: Participants] — Population: Caregiver-child dyads were enrolled in the trial. Data are presented for caregivers and children separately.
  Participants
    Caregivers: number analyzed (Participants) | 79 | 69 | 148
    Caregivers: <=18 years | 0 | 0 | 0
    Caregivers: Between 18 and 65 years | 79 | 68 | 147
    Caregivers: >=65 years | 0 | 1 | 1
    Children: number analyzed (Participants) | 79 | 69 | 148
    Children: <=18 years | 79 | 69 | 148
    Children: Between 18 and 65 years | 0 | 0 | 0
    Children: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Caregiver-child dyads were enrolled in the trial. Data are presented for caregivers and children separately.
  Years
    Caregivers: number analyzed (Participants) | 79 | 69 | 148
    Caregivers | 31.52 (6.83) | 32.52 (9.66) | 31.98 (8.26)
    Children: number analyzed (Participants) | 79 | 69 | 148
    Children | 2.71 (1.24) | 2.59 (1.22) | 2.66 (1.22)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Caregiver-child dyads were enrolled in the trial. Data are presented for caregivers and children separately.
  Participants
    Caregivers: number analyzed (Participants) | 79 | 69 | 148
    Caregivers: Female | 78 | 69 | 147
    Caregivers: Male | 1 | 0 | 1
    Children: number analyzed (Participants) | 79 | 69 | 148
    Children: Female | 40 | 34 | 74
    Children: Male | 39 | 35 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Caregiver-child dyads were enrolled in the trial. Data are presented for caregivers and children separately.
  Participants
    Caregivers: number analyzed (Participants) | 79 | 69 | 148
    Caregivers: Hispanic or Latino | 6 | 3 | 9
    Caregivers: Not Hispanic or Latino | 73 | 66 | 139
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
    Children: number analyzed (Participants) | 79 | 69 | 148
    Children: Hispanic or Latino | 6 | 2 | 8
    Children: Not Hispanic or Latino | 73 | 67 | 140
    Children: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Caregiver-child dyads were enrolled in the trial. Data are presented for caregivers and children separately.
  Participants
    Caregivers: number analyzed (Participants) | 79 | 69 | 148
    Caregivers: American Indian or Alaska Native | 0 | 0 | 0
    Caregivers: Asian | 0 | 0 | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 60 | 53 | 113
    Caregivers: White | 15 | 11 | 26
    Caregivers: More than one race | 1 | 4 | 5
    Caregivers: Unknown or Not Reported | 3 | 1 | 4
    Children: number analyzed (Participants) | 79 | 69 | 148
    Children: American Indian or Alaska Native | 0 | 0 | 0
    Children: Asian | 0 | 0 | 0
    Children: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Children: Black or African American | 61 | 55 | 116
    Children: White | 14 | 8 | 22
    Children: More than one race | 2 | 6 | 8
    Children: Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Weight of Mothers
Description: Body weight (kg) at baseline and follow-up assessments.
Time Frame: Baseline, 6 months, 12 months
Population: At 6-month visit, some participants unable to complete assessment due to COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Number analyzed (Participants) | 79 | 69
Kilograms
  Baseline | 88.65 (26.04) | 97.43 (31.29)
  6-months: number analyzed (Participants) | 54 | 66
  6-months | 85.96 (27.01) | 96.52 (28.97)
  12-months: number analyzed (Participants) | 70 | 63
  12-months | 85.94 (23.78) | 98.75 (30.77)

2. Primary Outcome: Weight of Children
Description: Body weight (kg) at baseline and follow-up assessments..
Time Frame: Baseline, 6 months, 12 months
Population: At 6-month visit, some participants unable to complete assessment due to COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Number analyzed (Participants) | 79 | 69
Kilograms
  Baseline | 13.88 (3.80) | 14.23 (5.10)
  6-months: number analyzed (Participants) | 53 | 66
  6-months | 15.40 (3.76) | 15.94 (5.21)
  12-months: number analyzed (Participants) | 70 | 63
  12-months | 16.83 (3.95) | 17.58 (5.80)

3. Secondary Outcome: Habit Strength of Targeted Behaviors
Description: Habit strength for caregivers will be assessed using the Self-Reported Habit Index (SRHI) specific to target behaviors on a scale from 1-5 with scores of 5 indicating higher caregiver habit strength for the target behavior.
Time Frame: Baseline, 6 months, 12 months
Population: At 6-month visit, some participants unable to complete assessment due to COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Number analyzed (Participants) | 79 | 69
Score on a scale
  Baseline- Fruit | 3.58 (0.96) | 3.67 (0.91)
  6-month- Fruit: number analyzed (Participants) | 54 | 65
  6-month- Fruit | 3.86 (0.81) | 3.95 (0.71)
  12-month- Fruit: number analyzed (Participants) | 71 | 62
  12-month- Fruit | 3.91 (0.96) | 4.26 (0.80)
  Baseline-Vegetables | 3.72 (1.00) | 3.79 (0.84)
  6-month-Vegetables: number analyzed (Participants) | 54 | 65
  6-month-Vegetables | 3.91 (0.82) | 4.07 (0.73)
  12-month-Vegetables: number analyzed (Participants) | 71 | 62
  12-month-Vegetables | 4.02 (1.01) | 4.18 (0.84)
  Baseline-Fried Food | 3.30 (1.09) | 2.99 (1.01)
  6-month-Fried Food: number analyzed (Participants) | 54 | 65
  6-month-Fried Food | 2.95 (1.09) | 2.89 (1.10)
  12-month-Fried Food: number analyzed (Participants) | 71 | 62
  12-month-Fried Food | 2.96 (1.07) | 3.13 (1.09)
  Baseline-SSB | 3.41 (1.14) | 3.13 (1.18)
  6-month-SSB: number analyzed (Participants) | 54 | 65
  6-month-SSB | 2.80 (1.13) | 2.98 (1.13)
  12-month-SSB: number analyzed (Participants) | 71 | 62
  12-month-SSB | 3.19 (1.22) | 3.27 (1.20)
  Baseline-Activity | 4.09 (0.83) | 3.99 (0.78)
  6-month-Activity: number analyzed (Participants) | 54 | 65
  6-month-Activity | 4.12 (0.73) | 4.08 (0.61)
  12-month-Activity: number analyzed (Participants) | 71 | 62
  12-month-Activity | 4.13 (0.78) | 4.29 (0.56)

4. Secondary Outcome: Household Environment Assessing the Number of Different Food Items Available
Description: Household environment assessing the number of different food items available in the home of the caregiver will be assessed using a modified Home Food Assessment (HFA) relating to the 4 food-related target behaviors (fruits, vegetables, sugary beverages, and fried foods). Higher values indicate more different food items in that category (fruits, vegetables, sugary beverages, and fried foods) are available within the home.
Time Frame: Baseline, 6 months, 12 months
Population: At 6-month visit, some participants unable to complete assessment due to COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: Available food items
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Number analyzed (Participants) | 79 | 69
Available food items
  Baseline-Fruit Availability | 5.01 (3.14) | 5.64 (3.75)
  6-month-Fruit Availability: number analyzed (Participants) | 54 | 65
  6-month-Fruit Availability | 6.00 (3.89) | 5.58 (3.40)
  12-month-Fruit Availability: number analyzed (Participants) | 71 | 62
  12-month-Fruit Availability | 5.28 (3.11) | 5.66 (2.72)
  Baseline-Vegetable Availability | 7.46 (3.66) | 7.29 (3.65)
  6-month-Vegetable Availability: number analyzed (Participants) | 54 | 65
  6-month-Vegetable Availability | 6.69 (4.01) | 7.89 (4.56)
  12-month-Vegetable Availability: number analyzed (Participants) | 71 | 62
  12-month-Vegetable Availability | 7.14 (3.83) | 7.34 (3.37)
  Baseline-Fried Food | 3.61 (3.05) | 3.30 (2.41)
  6-month-Fried Food: number analyzed (Participants) | 54 | 65
  6-month-Fried Food | 3.72 (2.65) | 3.71 (2.15)
  12-month-Fried Food: number analyzed (Participants) | 71 | 62
  12-month-Fried Food | 4.08 (2.68) | 3.71 (2.36)
  Baseline-SSB | 4.44 (2.89) | 3.84 (2.27)
  6-month-SSB: number analyzed (Participants) | 54 | 65
  6-month-SSB | 4.26 (2.66) | 4.09 (2.37)
  12-month-SSB: number analyzed (Participants) | 71 | 62
  12-month-SSB | 3.96 (2.43) | 3.68 (2.45)

5. Secondary Outcome: Household Environment Assessing the Number of Different Activity-promoting Items Available
Description: Household environment assessing the number of different activity-promoting items available in the home of the caregiver will be assessed using a modified Home - Inventory Describing Eating and Activity Development (H-IDEA) form. Higher values indicate more availability of different activity-promoting items in the home.
Time Frame: Baseline, 6 months, 12 months
Population: At 6-month visit, some participants unable to complete assessment due to COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: Available activity items
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Number analyzed (Participants) | 79 | 69
Available activity items
  Baseline | 3.96 (1.77) | 3.81 (1.58)
  6-month: number analyzed (Participants) | 54 | 65
  6-month | 4.59 (2.11) | 4.40 (2.15)
  12-month: number analyzed (Participants) | 71 | 62
  12-month | 4.30 (1.62) | 4.74 (2.17)

6. Other Pre Specified Outcome: Maternal Eating Practices
Description: Assessed using modified food and activity frequency measure from the National Health and Nutrition Examination Survey (NHANES), amended to measure target habit behaviors of feeding and activity. Scored on a scale from 0-6 with higher values indicated more frequent consumption of that food or engagement in that behavior.
Time Frame: Baseline, 6 months, 12 months
Population: At 6-month visit, some participants unable to complete assessment due to COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Number analyzed (Participants) | 79 | 69
Score on a scale
  Baseline-Fruit | 2.67 (1.73) | 2.33 (1.36)
  6-month-Fruit: number analyzed (Participants) | 54 | 65
  6-month-Fruit | 3.11 (1.68) | 2.57 (1.38)
  12-month-Fruit: number analyzed (Participants) | 71 | 62
  12-month-Fruit | 2.94 (1.76) | 2.94 (1.61)
  Baseline-Vegetable | 2.99 (1.42) | 2.49 (1.35)
  6-month-Vegetable: number analyzed (Participants) | 54 | 65
  6-month-Vegetable | 2.61 (1.42) | 2.66 (1.25)
  12-month-Vegetable: number analyzed (Participants) | 71 | 62
  12-month-Vegetable | 2.73 (1.49) | 2.84 (1.43)
  Baseline-Fried Food | 1.96 (1.46) | 1.23 (0.97)
  6-month-Fried Food: number analyzed (Participants) | 54 | 65
  6-month-Fried Food | 1.65 (1.29) | 1.37 (1.14)
  12-month-Fried Food: number analyzed (Participants) | 71 | 62
  12-month-Fried Food | 1.38 (1.09) | 1.35 (1.17)
  Baseline-Soda | 2.35 (2.04) | 1.72 (1.89)
  6-month-Soda: number analyzed (Participants) | 54 | 65
  6-month-Soda | 1.52 (1.44) | 1.48 (1.57)
  12-month-Soda: number analyzed (Participants) | 71 | 62
  12-month-Soda | 1.66 (1.71) | 1.77 (1.88)
  Baseline-Walk: number analyzed (Participants) | 79 | 68
  Baseline-Walk | 4.30 (1.84) | 4.16 (1.94)
  6-month-Walk: number analyzed (Participants) | 53 | 65
  6-month-Walk | 5.25 (1.52) | 4.78 (1.75)
  12-month-Walk: number analyzed (Participants) | 71 | 62
  12-month-Walk | 5.14 (1.53) | 4.95 (1.61)

7. Other Pre Specified Outcome: Maternal Feeding Practices
Description: Assessed using modified food and activity frequency measure from NHANES, amended to measure target habit behaviors of feeding and activity. Scored from 0-7 with higher values indicated more frequent consumption of food or engagement in the behavior.
Time Frame: Baseline, 6 months, 12 months
Population: At 6-month visit, some participants unable to complete assessment due to COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Number analyzed (Participants) | 79 | 69
Score on a scale
  Baseline-Fruit | 4.19 (1.96) | 4.14 (1.88)
  6-month-Fruit: number analyzed (Participants) | 54 | 65
  6-month-Fruit | 4.46 (1.73) | 4.54 (1.45)
  12-month-Fruit: number analyzed (Participants) | 71 | 62
  12-month-Fruit | 4.27 (1.65) | 4.37 (1.54)
  Baseline-Vegetable | 4.03 (1.87) | 3.70 (1.74)
  6-month-Vegetable: number analyzed (Participants) | 54 | 65
  6-month-Vegetable | 3.81 (1.69) | 4.02 (1.52)
  12-month-Vegetable: number analyzed (Participants) | 71 | 62
  12-month-Vegetable | 3.86 (1.55) | 3.77 (1.62)
  Baseline-Fried Food | 2.63 (1.70) | 2.13 (1.37)
  6-month-Fried Food: number analyzed (Participants) | 54 | 65
  6-month-Fried Food | 2.37 (1.14) | 2.29 (1.27)
  12-month-Fried Food: number analyzed (Participants) | 71 | 62
  12-month-Fried Food | 2.28 (1.24) | 2.11 (0.70)
  Baseline- Soda | 1.73 (1.64) | 1.46 (1.28)
  6-month-Soda: number analyzed (Participants) | 54 | 65
  6-month-Soda | 1.72 (1.35) | 1.68 (1.32)
  12-month-Soda: number analyzed (Participants) | 71 | 61
  12-month-Soda | 1.72 (1.22) | 1.85 (1.34)
  Baseline-Activity | 5.43 (1.89) | 5.22 (2.15)
  6-month-Activity: number analyzed (Participants) | 54 | 65
  6-month-Activity | 6.46 (1.18) | 6.09 (1.45)
  12-month-Activity: number analyzed (Participants) | 71 | 62
  12-month-Activity | 6.04 (1.61) | 5.92 (1.85)

8. Other Pre Specified Outcome: Caregiver Depressive Symptoms on the Personal Health Questionnaire Depression Scale (PHQ-8)
Description: The Personal Health Questionnaire Depression Scale (PHQ-8), a validated self-report measure of depressive symptoms experienced over the past two weeks, will be administered to caregivers. PHQ-8 scores range from 0-24, higher scores indicate higher caregiver depressive symptoms.
Time Frame: Baseline, 6 months, 12 months
Population: At 6-month visit, some participants unable to complete assessment due to COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Number analyzed (Participants) | 79 | 69
Score on a scale
  Baseline | 4.59 (4.19) | 4.42 (4.39)
  6-months: number analyzed (Participants) | 54 | 65
  6-months | 3.48 (3.64) | 3.08 (3.56)
  12-months: number analyzed (Participants) | 70 | 61
  12-months | 3.64 (3.56) | 3.03 (3.70)

9. Other Pre Specified Outcome: Number of Caregivers With Changes to Their Medical History
Description: Self-reported changes to medical history for caregivers (caregiver illnesses, etc.) will be collected.
Time Frame: 6 months, 12 months
Population: At 6-month visit, some participants unable to complete assessment due to COVID-19 pandemic.
Measure: Count of Participants; unit: Participants
Arm/Group | Home Visitation + HABITS Program | Standard Home Visitation Program
Number analyzed (Participants) | 71 | 65
Participants
  6-months: number analyzed (Participants) | 53 | 65
  6-months: Had a change to medical history in last 6-months | 2 | 4
  6-months: No change to medical history in last 6-months | 51 | 61
  12-months: number analyzed (Participants) | 71 | 62
  12-months: Had a change to medical history in last 6-months | 3 | 2
  12-months: No change to medical history in last 6-months | 68 | 60

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Home Visitation + HABITS Program: Caregivers; Home Visitation + HABITS Program: Children: The HABITS module will target 5 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, decreasing fried foods, and encouraging regular self-monitoring and self-weighing) aimed at reducing obesity risk in mothers or primary caregivers and children. Participants will receive the HABITS module in addition to their standard home visitation services.
  Home visitation + HABITS program: The HABITS program will target 5 key behaviors (physical activity, increasing fruit and vegetable consumption, decreasing sugary beverages, decreasing fried foods, and encouraging regular self-monitoring and self-weighing) aimed at reducing obesity risk in mothers or primary caregivers and children.
  Standard home visitation program: Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on promoting caregiver and child health by providing screenings and referrals, encouraging smoking cessation, promoting safe sleep practices, and strengthening children's school readiness and achievement, social/emotional and physical development.
- Standard Home Visitation Program: Caregivers; Standard Home Visitation Program: Children: Participants will receive the standard of care home visitation regularly delivered through the existing home visitation program without the HABITS module.
  Standard home visitation program: Treatment in the control arm includes the content and services typically provided by the home visitation partner, which is focused on promoting caregiver and child health by providing screenings and referrals, encouraging smoking cessation, promoting safe sleep practices, and strengthening children's school readiness and achievement, social/emotional and physical development.
Arm/Group | Home Visitation + HABITS Program: Caregivers | Home Visitation + HABITS Program: Children | Standard Home Visitation Program: Caregivers | Standard Home Visitation Program: Children
All-Cause Mortality (participants affected / at risk) | 0/79 | 1/79 | 1/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/79 | 1/79 | 1/69 | 0/69
Other Adverse Events (participants affected / at risk) | 0/79 | 0/79 | 0/69 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Visitation + HABITS Program: Caregivers (N=79) | Home Visitation + HABITS Program: Children (N=79) | Standard Home Visitation Program: Caregivers (N=69) | Standard Home Visitation Program: Children (N=69)
Hospitalization (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to COVID-19, there were protocol changes to the study and no data available for some of the 6-month study visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT03433456/Prot_SAP_ICF_000.pdf